CLINICAL TRIAL: NCT02423668
Title: Pseudophakic Anterior Chamber Depth Measurement in Second Eye Refinement Cataract Surgery
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Baixo Vouga (Other)
Responsible Party: Principal Investigator, Pedro Gil, MSc, MD, Centro Hospitalar do Baixo Vouga
Other Study IDs: CHBaixoVouga3
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cataract
Keywords: cataract surgery; biometry; second eye refinement; effective lens position
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 50% Partial adjustment: The prediction error for the first (PE1) and second (PE2) eyes was calculated as the difference between the observed post-operative refraction in spherical equivalent and the predicted post-operative refraction by the IOL Master for the implanted intra-ocular lens. This was obtained for the 3 formulae. Second eye refinement in the intra-ocular lens power selection for the second eye was performed using a theoretical 50% partial adjustment of the PE1. To relate refractive outcomes to pACD values, we performed subgroup analysis based in consecutive 50µm increments in inter-ocular asymmetry of pACD (50-600).
  Interventions: Procedure: 50% Partial adjustment
- No adjustment: The prediction error for the first (PE1) and second (PE2) eyes was calculated as the difference between the observed post-operative refraction in spherical equivalent and the predicted post-operative refraction by the IOL Master for the implanted intra-ocular lens. This was obtained for the 3 formulae. The intra-ocular lens power selection for the second eye was performed irrespective of the first eye prediction error. To relate refractive outcomes to pACD values, we performed subgroup analysis based in consecutive 50µm increments in inter-ocular asymmetry of pACD (50-600).
  Interventions: Procedure: No adjustment
- Full adjustment: The prediction error for the first (PE1) and second (PE2) eyes was calculated as the difference between the observed post-operative refraction in spherical equivalent and the predicted post-operative refraction by the IOL Master for the implanted intra-ocular lens. This was obtained for the 3 formulae. Second eye refinement in the intra-ocular lens power selection for the second eye was performed using a theoretical 100% partial adjustment of the PE1. To relate refractive outcomes to pACD values, we performed subgroup analysis based in consecutive 50µm increments in inter-ocular asymmetry of pACD (50-600).
  Interventions: Procedure: Full adjustment

INTERVENTIONS:
Procedure: 50% Partial adjustment — Second eye refinement in the IOL power selection for the second eye using a theoretical 50% partial adjustment of the PE1.
  Groups: 50% Partial adjustment
Procedure: No adjustment — IOL power selection for the second eye irrespective of first eye prediction error
  Groups: No adjustment
Procedure: Full adjustment — Second eye refinement in the IOL power selection for the second eye using a theoretical 100% partial adjustment of the PE1.
  Groups: Full adjustment

SUMMARY:
To study the effective lens position concept in second eye refinement (SER) cataract surgery, by relating inter-ocular symmetry of pseudophakic anterior chamber depth (pACD) measured in Pentacam and SER refractive outcomes.

DETAILED DESCRIPTION:
A retrospective chart review was conducted, including demographics (age and gender) and several parameters for both the first and second eyes, including the intra-ocular lens power calculation using the HofferQ, SRK/T and Holladay 1 formulas. Pentacam HR was used for pseudophakic anterior chamber depth measurement, and manual measurement was performed by a single investigator tracing a line between the anterior surface of the intra-ocular lens and the central corneal epithelium apex. Second eye refinement in the intra-ocular lens power selection for the second eye was performed using a theoretical 50% partial adjustment of the prediction error of the first eye. To relate refractive outcomes to pACD values, the investigators performed subgroup analysis based in consecutive 50µm increments in inter-ocular asymmetry of pACD (50-600).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for bilateral age-related cataract surgery

Exclusion Criteria:

* Age < 18 years old
* Previous or combined ocular surgery
* Manual extracapsular cataract extraction and not phacoemulsification
* Corneal sutures
* Implantation of any other IOL type
* IOL implanted in the sulcus
* Intra or postoperative complication
* Post-operative best-corrected visual acuity worse than 5/10
* Anterior corneal astigmatism>3.00 D
* Inadequate cooperation for Pentacam HR examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from the electronic database of a single ophthalmological center as having performed bilateral cataract surgery between 1st June 2013 and 24th July 2014
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Second eye mean absolute error | 4-6 weeks after second eye surgery
  Mean of the absolute value of the prediction error of the second eye

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gil, MSc, MD, Principal Investigator — Centro Hospitalar Baixo Vouga